CLINICAL TRIAL: NCT00057785
Title: A Phase II Study Of Intensity Modulated Radiation Therapy (IMRT) +/- Chemotherapy For Nasopharyngeal Cancer
Brief Title: Radiation Therapy With or Without Chemotherapy in Reducing Mouth Dryness in Patients With Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0225; CDR0000269314
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2016-12

CONDITIONS: Head and Neck Cancer; Oral Complications of Radiation Therapy; Radiation Toxicity
Keywords: oral complications of radiation therapy; radiation toxicity; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries | interventions — Cisplatin; Fluorouracil; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT +/- chemotherapy (Experimental): Intensity modulated radiation therapy (IMRT) for all patients and chemotherapy (cisplatin and fluorouracil) for patients with stage ≥ T2b and/or N+
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: Intensity modulated radiation therapy

INTERVENTIONS:
Drug: cisplatin — 100 mg/m^2 intravenously on days 1, 22, and 43 and 80 mg/m^2 intravenously on days 71, 99, and 127
Drug: fluorouracil — 1000 mg/m^2/day as 96-hour continuous infusion on days 71-74, 99-102, and 127-130
Radiation: Intensity modulated radiation therapy — The gross tumor and lymph node metastasis, Planning Target Volume (PTV) 70 (Clinical Target Volume [CTV] 70 with a 5 mm margin) will receive 70 Gy in 33 fractions at 2.12 Gy per fraction. Treatment will be delivered once daily, 5 fractions per week, over 6 weeks and 3 days.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy in different ways may cause less damage to normal tissue, prevent or lessen mouth dryness, and may help patients live more comfortably. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of specialized radiation therapy techniques with or without chemotherapy in reducing mouth dryness in patients who have nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the transportability of IMRT to a multi-institutional setting.
* Determine the rate of late xerostomia in patients with nasopharyngeal cancer treated with intensity-modulated radiotherapy (IMRT) with or without chemotherapy.
* Correlate reduction of side effects on salivary flow with compliance in patients treated with these regimens.
* Determine the rate of local-regional control, distant metastasis, and disease-free and overall survival of patients treated with these regimens.
* Determine the acute and late toxicity of these regimens in these patients.
* Determine chemotherapy compliance in patients treated with these regimens.

OUTLINE: Patients undergo daily intensity-modulated radiotherapy (IMRT) 5 days a week for approximately 6.5 weeks (total of 33 fractions) in the absence of disease progression or unacceptable toxicity.

Patients with stage T2b or greater and/or node-positive disease receive cisplatin IV over 20-30 minutes on days 1, 22, and 43 concurrently with IMRT followed by cisplatin IV over 20-30 minutes and fluorouracil IV over 96 hours starting on days 71, 99, and 127.

Quality of life is assessed through saliva measurement at baseline and then at 3, 6, and 12 months after IMRT.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 64 patients will be accrued for this study within 36-40 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-IVB squamous cell carcinoma of the nasopharynx

  * WHO I-III
  * No stage IVC disease
  * No evidence of distant metastasis
* Measurable or evaluable disease
* Must have been treated with primary radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* White blood cell count (WBC) at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine no greater than 1.6 mg/dL
* Creatinine clearance at least 60 mL/min

Other

* Not pregnant (If stage T2b or greater or node-positive disease)
* Negative pregnancy test (If stage T2b or greater or node-positive disease)
* No other prior head and neck cancer
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No active untreated infection
* No other major medical or psychiatric illness that would preclude study entry
* Nutritional and general physical condition compatible with radiotherapy NOTE: *If stage T2b or greater or node-positive disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 6 months since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 6 months since prior radiotherapy for head and neck cancer

Surgery

* No prior head and neck surgery to the primary tumor or lymph nodes except incisional or excisional biopsies

Other

* No other concurrent experimental therapy for cancer
* No amifostine or pilocarpine during or for 3 months after radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-02; Primary Completion 2007-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (17):
- United States (17):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Davis Cancer Center, Davis, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Albuquerque Regional Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - Akron City Hospital, Akron, Ohio
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - McKay-Dee Hospital Center, Ogden, Utah
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Chen A, Lee N, Yang C, Liu T, Narayan S, Vijayakumar S, Purdy J. Comparison of intensity-modulated radiotherapy using helical tomotherapy and segmental multileaf collimator-based techniques for nasopharyngeal carcinoma: dosimetric analysis incorporating quality assurance guidelines from RTOG 0225. Technol Cancer Res Treat. 2010 Jun;9(3):291-8. doi: 10.1177/153303461000900308. PMID 20441239
- [Result] Lee N, Harris J, Garden AS, Straube W, Glisson B, Xia P, Bosch W, Morrison WH, Quivey J, Thorstad W, Jones C, Ang KK. Intensity-modulated radiation therapy with or without chemotherapy for nasopharyngeal carcinoma: radiation therapy oncology group phase II trial 0225. J Clin Oncol. 2009 Aug 1;27(22):3684-90. doi: 10.1200/JCO.2008.19.9109. Epub 2009 Jun 29. PMID 19564532
- [Result] Lee NY, Harris J, Garden A, et al.: Phase II multi-institutional study of IMRT ± chemotherapy for nasopharyngeal carcinoma (RTOG 0225): preliminary results. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-23, S13-14, 2007.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMRT +/- Chemotherapy
Started | 68
Completed | 68 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | IMRT +/- Chemotherapy
Number analyzed (Participants) | 68
Age, Continuous [Median (Full Range); unit: years] | 48.5 [18 to 73]
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Protocol Compliance of Intensity-modulated Radiotherapy Treatment Delivered
Description: Patients scored by the study chairs as no variation or minor variation were considered compliant, while patients scored as major variation or inevaluable were considered non-compliant. The number being reported is the number non-compliant. A compliance rate of 90% was targeted with 75% or lower being considered unacceptable. Fifty-seven patients were required with types I and II error rates both 0.10. If 10 or more patients out of 57 were non-compliant, the treatment would be unacceptable, per a two-stage Fleming multiple testing procedure.
Time Frame: From start of treatment to end of treatment
Population: First 57 eligible patients who started study treatment.
Measure: Number; unit: participants
Arm/Group | IMRT +/- Chemotherapy
Number analyzed (Participants) | 57
participants | 9

2. Secondary Outcome: Rate of Xerostomia at 1 Year (Grade ≥ 2)
Time Frame: From start of treatment to 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Locoregional Control at 2 Years
Time Frame: From registration to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Whole Mouth Saliva Output Relative to Pretreatment Measurements
Time Frame: From start of treatment to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Other Acute and Late Toxicities
Time Frame: From start of treatment to last follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Chemotherapy Compliance
Time Frame: From start of treatment to end of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for nonserious adverse events (AE).
Arm/Group | IMRT +/- Chemotherapy
Serious Adverse Events (participants affected / at risk) | 55/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT +/- Chemotherapy (N=68)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Hemoglobin decreased (Blood and lymphatic system disorders) | 10
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 4
Edema NOS (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular arrhythmia NOS (Cardiac disorders) | 1
Ventricular arrhythmia NOS (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 8
Hearing-Other (Ear and labyrinth disorders) | 3
Otitis externa (exc boil of meatus) NOS (Ear and labyrinth disorders) | 2
Endocrine-Other (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Diarrhea NOS (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 16
Esophageal spasm (Gastrointestinal disorders) | 6
Esophagitis NOS (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 21
Radiation mucositis (Gastrointestinal disorders) | 28
Salivary gland disorder NOS (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 6
Vomiting NOS (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 6
Pain due to radiation (General disorders) | 6
Pain-other (General disorders) | 6
Pyrexia (General disorders) | 1
Implant infection (Infections and infestations) | 1
Infection NOS (Infections and infestations) | 3
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 4
Infection with unknown ANC (Infections and infestations) | 1
Infection, Other (Infections and infestations) | 2
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
CD4 lymphocytes decreased (Investigations) | 1
Inappropriate ADH secretion (Investigations) | 1
Leukocytes for BMT (Investigations) | 1
Leukopenia NOS (Investigations) | 4
Lymphopenia (Investigations) | 11
Neutropenia (Investigations) | 20
Platelet count decreased (Investigations) | 4
Weight decreased (Investigations) | 12
Weight increased (Investigations) | 1
Acidosis NOS (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Blood albumin decreased (Metabolism and nutrition disorders) | 2
Blood magnesium decreased (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 11
Hyperglycemia NOS (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache NOS (Nervous system disorders) | 1
Neurologic-Other (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Anxiety NEC (Psychiatric disorders) | 1
Depression NEC (Psychiatric disorders) | 1
Hallucination NOS (Psychiatric disorders) | 2
Renal failure NOS (Renal and urinary disorders) | 1
Renal/GU-Other (Renal and urinary disorders) | 2
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Skin-Other (Skin and subcutaneous tissue disorders) | 2
Hemorrhage NOS (Vascular disorders) | 1
Hypotension NOS (Vascular disorders) | 6
Thrombosis NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT +/- Chemotherapy (N=68)
Hematologic-Other (Blood and lymphatic system disorders) | 8
Hemoglobin decreased (Blood and lymphatic system disorders) | 51
Edema NOS (Cardiac disorders) | 13
Earache (Ear and labyrinth disorders) | 4
Hearing impaired (Ear and labyrinth disorders) | 33
Hearing-Other (Ear and labyrinth disorders) | 17
Late RT toxicity: Auditory/hearing: NOS (Ear and labyrinth disorders) | 32
Otitis media serous NOS (Ear and labyrinth disorders) | 7
Hypothyroidism (Endocrine disorders) | 10
Constipation (Gastrointestinal disorders) | 14
Diarrhea NOS (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 61
Dysphagia (Gastrointestinal disorders) | 24
Esophagitis NOS (Gastrointestinal disorders) | 28
GI-other (Gastrointestinal disorders) | 8
Late RT toxicity: Esophagus: NOS (Gastrointestinal disorders) | 28
Late RT toxicity: Larynx: NOS (Gastrointestinal disorders) | 13
Late RT toxicity: Mucous membrane: NOS (Gastrointestinal disorders) | 41
Late RT toxicity: Salivary gland: NOS (Gastrointestinal disorders) | 51
Nausea (Gastrointestinal disorders) | 46
Radiation mucositis (Gastrointestinal disorders) | 50
Salivary gland disorder NOS (Gastrointestinal disorders) | 59
Stomatitis (Gastrointestinal disorders) | 15
Vomiting NOS (Gastrointestinal disorders) | 31
Fatigue (General disorders) | 50
Late RT toxicity: Other: NOS (General disorders) | 33
Pain due to radiation (General disorders) | 24
Pain-other (General disorders) | 24
Pyrexia (General disorders) | 10
Rigors (General disorders) | 5
Infection NOS (Infections and infestations) | 7
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 43
Late RT toxicity: Skin (within RT field): NOS (Injury, poisoning and procedural complications) | 22
Late RT toxicity: Subcutaneous tissue (within RT field): NOS (Injury, poisoning and procedural complications) | 27
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 9
Blood alkaline phosphatase NOS increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 6
Blood creatinine increased (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 5
Leukopenia NOS (Investigations) | 50
Lymphopenia (Investigations) | 16
Metabolic-Other (Investigations) | 7
Neutropenia (Investigations) | 33
Platelet count decreased (Investigations) | 18
Weight decreased (Investigations) | 40
Anorexia (Metabolism and nutrition disorders) | 18
Blood albumin decreased (Metabolism and nutrition disorders) | 19
Blood magnesium decreased (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 19
Hyperglycemia NOS (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 17
Hypokalemia (Metabolism and nutrition disorders) | 15
Hyponatremia (Metabolism and nutrition disorders) | 26
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Joint, muscle, or bone-Other (Musculoskeletal and connective tissue disorders) | 4
Late RT toxicity: Bone (incl. osteonecrosis): NOS (Musculoskeletal and connective tissue disorders) | 4
Late RT toxicity: Joint: NOS (Musculoskeletal and connective tissue disorders) | 13
Dizziness (exc vertigo) (Nervous system disorders) | 4
Headache NOS (Nervous system disorders) | 10
Neuralgia NOS (Nervous system disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 23
Taste disturbance (Nervous system disorders) | 19
Confusion (Psychiatric disorders) | 4
Insomnia NEC (Psychiatric disorders) | 4
Renal/GU-Other (Renal and urinary disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 20
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6
Skin discoloration (Skin and subcutaneous tissue disorders) | 9
Skin-Other (Skin and subcutaneous tissue disorders) | 8
Toxicoderma (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.